CLINICAL TRIAL: NCT03340194
Title: Evaluation of Calcinosis Prevalence in Systemic Sclerosis : a Cross Sectional Study Evaluating Calcinosis Cutis Prevalence by Hand and Feet Radiographic Assessment in Systemic Sclerosis Patients and Study Their Correlation With Organ Injury
Brief Title: Evaluation of Calcinosis in Systemic Sclerosis
Acronym: CALCIDERMIS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016_43; 2017-A01822-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; Calcinosis cutis
MeSH Terms: conditions — Scleroderma, Systemic; Calcinosis Cutis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Systemic sclerosis patients
  Interventions: Radiation: Radiography; Procedure: Veinous punction

INTERVENTIONS:
Radiation: Radiography — Radiography of the hand and feet (face incident) the day of the inclusion
Procedure: Veinous punction — Blood sample to analysis VEGF, endothelin 1, endostatin and P/GF, (ELISA method)

SUMMARY:
Systemic sclerosis is a rare pathology characterized by fibrosis and vascular lesion with skin, pulmonary, digestive and cardiac localisation. Calcinosis cutis is commonly described, but its prevalence and appear few documented in literature. Moreover, this studies used clinical observation to determine presence or absence of calcification, and rarely radiography, in particular for feet localisation. In the same way, skin calcification and organ injury association appear unclear. The aim of the study is firstly to determine prevalence of calcinosis cutis, with hand and feet radiography realisation in a cohort of systemic sclerosis patient. Secondly, will be determine the correlation between calcinosis and organ injury.

ELIGIBILITY:
Inclusion Criteria:

* Systemic sclerosis presenting ACR-EULAR 2013 criteria
* Given their consent
* Titulary of health insurance

Exclusion Criteria:

* Dermatomyositis overlap
* Pregnant or breastfeeding women
* Imprisoned person
* Refuse of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systemic sclerosis patient in the national reference center for scleroderma (Lille, France)
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Calcinosis cutis prevalence by radiographic assessment | at inclusion ( baseline)

SECONDARY OUTCOMES:
Demographic data | at inclusion ( baseline)
Rodnan score | at inclusion ( baseline)
Visceral localisation evaluation (cardiac, pulmonary, digestive) | at inclusion ( baseline)
EUSTAR score | at inclusion ( baseline)
Medsger score | at inclusion ( baseline)
Quality of life evaluation (HAQ modified questionary) | at inclusion ( baseline)
Biologic vascular markers : VEGF, endothelin 1, endostatin and P/GF, (ELISA method) | at inclusion ( baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent SOBANSKI, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France